CLINICAL TRIAL: NCT01430377
Title: Side Branch Predilatation Strategy in Coronary Bifurcation Lesion Stenting (SBPS)
Acronym: SBPS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medica Cor Heart Hospital (Other)
Responsible Party: Principal Investigator, Dobrin Vassilev MD, PhD, Dobrin Vassilev MD, PhD, Medica Cor Heart Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBPS
Record Dates: First submitted 2011-09-03; First posted 2011-09-08 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Coronary Ostium Stenosis; Myonecrosis
Keywords: periprocedural myonecrosis; procedure time; fluoroscopy time

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SB predilatation (Experimental)
  Interventions: Procedure: SB predilatation; Procedure: No SB predilatation

INTERVENTIONS:
Procedure: SB predilatation — Initial SB [predilatation.
Procedure: No SB predilatation — Without SB predilatation

SUMMARY:
The role of Side Branch (SB) predilatation during coronary bifurcation lesion percutaneous coronary intervention (PCI) is still not established. The predilatation could potentially damage SB ostium by vessel dissection, making subsequent wiring problematic. However, predilatation could eliminate SB ostial stenosis obviating need for further SB treatment after main vessel stent implantation. The aim of the study is to assess in random fashion the periprocedural myonecrosis, complication rates and time for SB rewiring in groups with and without SB predilatation.

ELIGIBILITY:
1. Inclusion Criteria

   * Subject at least 18 years of age.
   * Subject able to verbally confirm understandings of risks, benefits of receiving PCI for true bifurcation lesions, and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
   * Target main branch lesion(s) located in a native coronary artery with diameter of ≥ 2.5 mm and ≤ 4.5 mm. Target side branch lesion(s) located in a native coronary artery with diameter of ≥ 2.0 mm.
   * Target lesion(s) amenable for PCI with balloon angioplasty of the side branch.
2. Exclusion Criteria

   * ST-segment elevation myocardial infarction (STEMI)
   * Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
   * Subjects who refuse to give informed consent.
   * Subjects with left ventricle ejection fraction <30%
   * Subjects with moderate or severe degree valvular heart disease or primary cardiomyopathy
   * Contraindications for 12 months double antiplatelet therapy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-04 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Time for rewiring SB | 24h

SECONDARY OUTCOMES:
Periprocedural myonecrosis | 24 h
MACE | 12 months
  death, MI, TVR

CONTACTS AND LOCATIONS:
Locations (1):
- Medica Cor Heart Hospital, Rousse, Bulgaria